CLINICAL TRIAL: NCT04396587
Title: Non-analgesic Effects Produced by Equipotent Analgesic Doses of Sufentanil, Hydromorphone, and Oxycodone in Female Patients Before Anesthesia Induction
Brief Title: Non-analgesic Effects Produced by Equipotent Analgesic Doses of Sufentanil, Hydromorphone, and Oxycodone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yanqi, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAESHO
Record Dates: First submitted 2020-05-16; First posted 2020-05-20 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Opioid Use
MeSH Terms: interventions — Sufentanil; Hydromorphone; Oxycodone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sufentanil (Experimental): Sufentanil(0.1μg/kg)
  Interventions: Drug: Sufentanil
- Hydromorphone (Experimental): Hydromorphone(20μg/kg）
  Interventions: Drug: Hydromorphone
- Oxycodone (Experimental): Oxycodone(60μg/kg)
  Interventions: Drug: Oxycodone
- normal saline (Placebo Comparator): 10ml
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Sufentanil — Sufentanil(0.1μg/kg) was administered before anesthesia induction.
  Arms: Sufentanil
Drug: Hydromorphone — Hydromorphone(20μg/kg)was administered before anesthesia induction.
  Arms: Hydromorphone
Drug: Oxycodone — Oxycodone(60μg/kg) was administered before anesthesia induction.
  Arms: Oxycodone
Drug: normal Saline — normal saline 10ml
  Arms: normal saline

SUMMARY:
This study aimed to investigate Non-analgesic Effects Produced by Equipotent Analgesic Doses of Sufentanil, Hydromorphone, and Oxycodone in female patients. Methods: A total of 60 patients were randomly divided into 4 groups, with 20 patients in each group. Sufentanil(0.1μg/kg), Hydromorphone(20μg/kg), or Oxycodone(60μg/kg) ,saline(10ml)was administered before anesthesia induction. Bispectral Index (BIS), Respiratory rate(RR), other non-analgesic effects at Tb (entering room), T0 (drug administration), T1 (2min), T2 (4min), T3(6min), T4(8min), T5(10min), T6(20min) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists GradeⅠ-II;
* Patients undergo low-risk elective surgery for benign diseases (including laparoscopic ovarian cyst removal, laparoscopic tubal ligation, laparoscopic tubal drainage, breast operation, thyroid operation, etc) ;
* Aged 18-45 years;
* Body Mass Index 18-25kg/m2, weight 40-65 kilograms;
* Agreed to participate in the research

Exclusion Criteria:

* Difficult airway;
* upper respiratory tract infection within 2 weeks;
* history of allergy or long-term use of propofol and opioids;
* self-rating anxiety scale before operation indicates anxiety;
* pregnancy or lactation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Respiratory rate | 20 minutes after administration
  Number of breaths per minute
Bispectral Index | 20 minutes after administration
  bispectral index(BIS): assessing the sedation, placed on the patient's forehead, BIS values 0-100, and the higher score means patients are more conscious
dizziness | 20 minutes after administration
  a temporary feeling that your sense of balance is not good and that you may fall down

SECONDARY OUTCOMES:
itch | 20 minutes after administration
  itch
nausea or vomiting | 20 minutes after administration
  nausea or vomiting
drowsiness | 20 minutes after administration
  drowsiness
sweating | 20 minutes after administration
  sweating

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No